CLINICAL TRIAL: NCT01720472
Title: Implementing a Physical and Cognitive Performance Assessment Cohort in the MURDOCK Study Community Registry and Biorepository
Acronym: PPS
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00036608
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Aging; Physical Functioning; Cognitive Functioning; Fitness
Keywords: Aging; Healthy Aging; Physical Performance; Physical Functioning; Cognitive Functioning; Fitness; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Serum and plasma samples collected from MURDOCK Study enrollment visit and two year follow up Physical Performance visit.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Community, Physical Performance
  Interventions: Genetic: Biomarker studies

INTERVENTIONS:
Genetic: Biomarker studies

SUMMARY:
The purpose of this study is to use the MURDOCK Horizon 1.5 infrastructure (Duke Instutional Review Board Pro00011196) to specifically target and enroll 1,000 participants across age groups and other demographic categories in order to develop a diverse cohort with specific physical and cognitive performance data paired with biological samples.

DETAILED DESCRIPTION:
The MURDOCK Study, proposes this Horizon 2 study to collect a brief physical and cognitive performance assessment from 1,000 MURDOCK Registry participants. Blood sample aliquots will also be obtained. These physical and cognitive performance data, paired with -omics data from plasma and serum sample analyses, offer promise in the discovery of biomarkers for functional decline. This research will provide an important basis for our understanding of the physical, lifestyle, and genetic factors which, over the lifespan, contribute to changes in physical and cognitive capabilities as we age.

ELIGIBILITY:
Inclusion Criteria:

* A resident of Cabarrus County and/or the city of Kannapolis (and surrounding regions) or certain portions of Rowan, Mecklenburg, or Stanly counties in North Carolina for 6 or more months of the year.
* Age 30 or older

Exclusion Criteria:

* Female that is currently pregnant
* Having had a heart attack, angina, congestive heart failure, or fluid in the lungs within the past 6 months
* Participant that requires consent by a legally authorized representative
* Participant that cannot walk 30ft without human assistance

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include 1,000 participants ages 30 and older living in Cabarrus County and/or the city of Kannapolis, or certain portions of Rowan, Mecklenburg, or Stanly counties in North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-05; Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Implementing a Physical and Cognitive Performance Assessment Cohort in the MURDOCK Study Community Registry and Biorepository | Upto 2 years or 24 months
  Factors associated with physical function and physical activity and change in physical activity and function over two-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam C Morey, Ph.D., Principal Investigator — Duke University
Locations (6):
- United States (6):
  - Bethesda Health Center, Charlotte, North Carolina
  - McGill Family Medicine, Concord, North Carolina
  - Carolinas Medical Center NorthEast Medical Arts Building, Concord, North Carolina
  - Ada Jenkins Center, Davidson, North Carolina
  - Harrisburg Sleep Center, Harrisburg, North Carolina
  - Lake Norman Community Health Clinic, Huntersville, North Carolina

REFERENCES:
- [Derived] Parker D, Sloane R, Pieper CF, Hall KS, Kraus VB, Kraus WE, Huebner JL, Ilkayeva OR, Bain JR, Newby LK, Cohen HJ, Morey MC. Age-Related Adverse Inflammatory and Metabolic Changes Begin Early in Adulthood. J Gerontol A Biol Sci Med Sci. 2019 Feb 15;74(3):283-289. doi: 10.1093/gerona/gly121. PMID 29985987
- See also: MURDOCK Study Physical Performance Cohort — http://www.murdock-study.com/